CLINICAL TRIAL: NCT03505736
Title: The ESPRIT Study: Estrogen Suppression and Perfusion Reserve With Aromatase-Inhibitor Treatment in Premenopausal Women With Breast Cancer
Brief Title: Stress Test in Detecting Heart Damage in Premenopausal Women With Stage I-III Breast Cancer
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB00049171; NCI-2018-00588 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CCCWFU 98118 (Other: Wake Forest University Health Sciences); P30CA012197 (NIH)
Record Dates: First submitted 2018-04-12; First posted 2018-04-23 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Anatomic Stage I Breast Cancer AJCC v8; Anatomic Stage IA Breast Cancer AJCC v8; Anatomic Stage IB Breast Cancer AJCC v8; Anatomic Stage II Breast Cancer AJCC v8; Anatomic Stage IIA Breast Cancer AJCC v8; Anatomic Stage IIB Breast Cancer AJCC v8; Anatomic Stage III Breast Cancer AJCC v8; Anatomic Stage IIIA Breast Cancer AJCC v8; Anatomic Stage IIIB Breast Cancer AJCC v8; Anatomic Stage IIIC Breast Cancer AJCC v8; Premenopausal; Prognostic Stage I Breast Cancer AJCC v8; Prognostic Stage IA Breast Cancer AJCC v8; Prognostic Stage IB Breast Cancer AJCC v8; Prognostic Stage II Breast Cancer AJCC v8; Prognostic Stage IIA Breast Cancer AJCC v8; Prognostic Stage IIB Breast Cancer AJCC v8; Prognostic Stage III Breast Cancer AJCC v8; Prognostic Stage IIIA Breast Cancer AJCC v8; Prognostic Stage IIIB Breast Cancer AJCC v8; Prognostic Stage IIIC Breast Cancer AJCC v8
MeSH Terms: interventions — Adenosine; Magnetic Resonance Spectroscopy; regadenoson

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Diagnostic (stress test): Within 2 years of initiating anti-estrogen therapy or 2 years after completing chemotherapy, participants undergo a stress test which consists of receiving adenosine IV over 1-5 minutes or regadenoson IV over 2 minutes and then undergoing CMR imaging over 45-60 minutes at baseline, and again 3-6 months later.
  Interventions: Biological: Adenosine; Procedure: Magnetic Resonance Imaging; Drug: Regadenoson; Procedure: Stress Management Therapy

INTERVENTIONS:
Biological: Adenosine — Given IV
Procedure: Magnetic Resonance Imaging — Undergo CMR imaging
  Other Names: Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MRI; MRI Scan; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging
Drug: Regadenoson — Given IV
  Other Names: CVT-3146
Procedure: Stress Management Therapy — Undergo stress test

SUMMARY:
This pilot trial studies how well a stress test works in detecting heart damage in premenopausal women with stage I-III breast cancer. Giving a stress test with adenosine or regadenoson and cardiovascular magnetic resonance imaging may help doctors detect heart damage caused by breast cancer treatments including chemotherapy and aromatase inhibitors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To describe decrements in left ventricular myocardial microcirculatory perfusion reserve in premenopausal women treated with an aromatase inhibitor for high-risk hormone receptor-positive breast cancer and in premenopausal women treated without an aromatase inhibitor for triple negative breast cancer over three to six months of in the first 24 months on an aromatase inhibitor or after cessation of chemotherapy, respectively.

SECONDARY OBJECTIVES:

I. To describe changes between the cohorts with hormone receptor-positive and triple negative breast cancer in other measures of cardiovascular function as measured by myocardial rest T1 (myocardial fibrosis burden) and left ventricular ejection fraction (LVEF) measured noninvasively with cardiovascular magnetic resonance (CMR) imaging over three to six months.

II. To describe the relationship of clinical and demographic variables in relation to their potential contribution to changes in left ventricular myocardial microcirculatory perfusion reserve over three to six months in both groups.

III. To study the overall feasibility of accruing and retaining premenopausal women with stage I-III breast cancer in a trial using adenosine stress CMR to assess myocardial perfusion reserve (MPR) and other parameters of cardiovascular health.

OUTLINE:

Within 2 years of initiating anti-estrogen therapy or 2 years after completing chemotherapy, participants undergo a stress test which consists of receiving adenosine intravenously (IV) over 1-5 minutes or regadenoson IV over 2 minutes and then undergoing CMR imaging over 45-60 minutes at baseline and then 3-6 months later.

After completion of study, participants are followed up at 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Women who were premenopausal at the time of breast cancer diagnosis; (premenopausal is defined as per National Comprehensive Cancer Network (NCCN) criteria
* Breast cancer treatment is within three years of initiating anti-estrogen therapy and includes medically or surgically induced menopause (HR-positive tumor) or three years of completing chemotherapy (HR-negative tumor)
* Diagnosed with stage I-III breast cancer OR with metastatic breast cancer and receiving ovarian suppression function and aromatase inhibitors as their first non-chemotherapy regimen in the metastatic setting (can include CDK inhibitor with aromatase inhibitor)
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Ability to understand and the willingness to sign an Institutional Review Board (IRB)-approved informed consent document (either directly or via a legally authorized representative)

Exclusion Criteria:

* Women with human epidermal growth factor-2 (HER2) positive breast cancer would be excluded from this pilot given the confounding issue of the cardiotoxicity associated with HER2-directed therapies.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to adenosine (or regadenoson for those with history of asthma or chronic obstructive pulmonary disease [COPD])
* Those with contraindications for MRI such as some breast expanders, ferromagnetic cerebral aneurysm clips or other intracranial metal, pacemakers, defibrillators, functioning neurostimulator devices or other implanted electronic devices
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study; a pregnancy test is required, unless the patient has undergone either a bilateral oophorectomy, hysterectomy or both
* Coronary revascularization in the past 6 months or known severe multi-vessel coronary artery disease (CAD) previously determined to be not amenable to mechanical intervention
* Ongoing, unrelieved symptoms thought to represent cardiac ischemia and requiring immediate cardiac catheterization

Max Age: 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Adults with stage I-III breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2018-06-21 (Actual); Primary Completion 2020-03-05 (Actual); Study Completion 2020-03-05 (Actual)

PRIMARY OUTCOMES:
Myocardial perfusion reserve index (MPRI) | Baseline and 3-6 months
  Will first estimate 95% confidence intervals for each group at each time point as well as for the change from baseline to 3-6-months in each group.

SECONDARY OUTCOMES:
Myocardial rest myocardial fibrosis burden (T1) and left ventricular ejection fraction (LVEF) | Baseline and 3-6 months
  Will be used to correlate myocardial perfusion with T1 and myocardial function (LVEF).
Change in MPRI measures | Baseline to 3-6 months
  Change in MPRI measures (overall and within each group) will be compared using 2-sample t-tests for binary variables. Correlations will be estimated between BMI and the change in MPRI measures.
Accrual rate defined as based on the number of patients who participate compared to the total number of patients approached | Baseline and 3-6 months
  Will capture data for those approached and consenting or declining and any reasons given for declining participation into the study. Will be assessed by estimating counts and percent's and corresponding 95% Clopper-Pearson exact binomial confidence intervals. Will be compared to the total number of patients enrolled.
Retention rate defined the number of patients who are enrolled and complete both assessments | Baseline and 3-6 months
  Will be assessed by estimating counts and percent's and corresponding 95% Clopper-Pearson exact binomial confidence intervals. Will be compared to the total number of patients enrolled.

CONTACTS AND LOCATIONS:
Overall Officials: Emily Douglas, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States